CLINICAL TRIAL: NCT03135028
Title: A Phase 1b Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Entospletinib (ENTO) as Monotherapy in Japanese Subjects With Relapsed or Refractory Hematologic Malignancies and in Combination With Chemotherapy in Japanese Subjects With Previously Untreated Acute Myeloid Leukemia (AML)
Brief Title: Entospletinib (ENTO) as Monotherapy and in Combination With Chemotherapy in Japanese Adults
Acronym: Japanese AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No signal of efficacy with Entospletinib
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-429-4104
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Hematologic Malignancy; Acute Myeloid Leukemia
Keywords: Relapsed or Refractory Hematologic Malignancy; Previously untreated AML
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Recurrence | interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ENTO monotherapy (Group A) (Experimental): Participants with relapsed or refractory hematologic malignancies will receive ENTO twice daily of every 28-day cycle until participants meet treatment discontinuation criteria or do not experience clinical benefit.
  Interventions: Drug: Entospletinib
- ENTO + cytarabine + daunorubicin (Group B) (Experimental): Lead-in (Cycle 0): Participants with previously untreated AML will receive ENTO twice daily for 14 days.
  Induction (Up to 2 cycles): ENTO in combination with daunorubicin and cytarabine for up to two 28-day cycles.
  Post-remission chemotherapy (at least 2 cycles, up to 4 cycles): Some participants (who have achieved complete remission [CR] or morphologic complete remission with incomplete blood count recovery [CRi] and do not require or cannot proceed to allogeneic stem cell transplantation [SCT] and participants who are awaiting a donor or transitioning to allogeneic SCT per investigator discretion) will have the option to receive post-remission chemotherapy with ENTO twice daily in combination with high-dose cytarabine (Hi-DAC) for up to four 28-day cycles.
  Interventions: Drug: Entospletinib; Drug: Daunorubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Entospletinib — 400 mg (2 × 200 mg tablets) orally twice daily
  Other Names: GS-9973; ENTO
Drug: Daunorubicin — 60 mg/m^2 administered intravenously daily on Days 1 to 3 of each 28-day induction cycle
  Arms: ENTO + cytarabine + daunorubicin (Group B)
Drug: Cytarabine — 100 mg/m^2 intravenous administration twice daily on Days 1 to 7 of each 28-day induction cycle
  Hi-DAC: 3 g/m^2 IV administration twice daily on days 1, 3, and 5 (≤ 60 years of age) or 1 g/m^2 IV administration once daily on Days 1 to 5 (> 60 years of age) of each 28-day post-remission cycle
  Arms: ENTO + cytarabine + daunorubicin (Group B)

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of entospletinib (ENTO) monotherapy and in combination with chemotherapy in Japanese participants.

ELIGIBILITY:
Key Inclusion Criteria:

* ENTO monotherapy (Group A): relapsed or refractory hematologic malignancies by World Health Organisation (WHO) criteria and who are not eligible to receive standard of care
* ENTO + cytarabine + daunorubicin (Group B): previously untreated AML by WHO criteria, who are deemed fit for cytarabine and daunorubicin (7+3) induction chemotherapy and are able to undergo up to 2 cycles of induction chemotherapy, as determined by the treating physician
* Must have been born in Japan and must not have lived outside of Japan for a period > 1 year in the 5 years prior to Day 1 of study treatment
* Must be able to confirm the Japanese origin of their maternal and paternal ancestry

Key Exclusion Criteria:

* Known active central nervous system or leptomeningeal leukemic involvement
* Ongoing liver injury, or known infection with chronic active hepatitis C virus (HCV) or chronic active hepatitis B virus (HBV)

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- Japan (6):
  - University of Fukui Hospital, Fukui
  - Kyushu University Hospital, Fukuoka
  - Tokai University Hospital, Kanagawa
  - Tohoku University Hospital, Miyagi
  - Kindai University Hospital, Ōsaka
  - NTT Medical Center Tokyo, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Japan. The first participant was screened on 19 May 2017. The last study visit occurred on 26 February 2019.
Pre-assignment Details: 13 participants were screened.
Groups:
- ENTO 400 mg: Participants received entospletinib (ENTO) 400 mg (2 × 200 mg tablets) orally twice daily in a fasted state on Days 1 through 28 of every 28-day cycle, and continued on study treatment as long as the participant experienced benefit and did not meet the criteria for study treatment discontinuation.
Period: Overall Study
Arm/Group | ENTO 400 mg
Started | 9
Completed | 0
Not Completed | 9
Not completed — Death | 6
Not completed — Study Terminated by Sponsor | 2
Not completed — Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who received at least 1 dose of study drug (ENTO).
Groups:
- ENTO 400 mg: Participants received ENTO 400 mg (2 × 200 mg tablets) orally twice daily in a fasted state on Days 1 through 28 of every 28-day cycle, and continued on study treatment as long as the participant experienced benefit and did not meet the criteria for study treatment discontinuation.
Arm/Group | ENTO 400 mg
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 8
  Race: Black | 0
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: White | 0
  Race: Not Permitted | 0
  Race: Other | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0
  Ethnicity: Not Hispanic or Latino | 9
  Ethnicity: Not Permitted | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Laboratory Abnormalities Defined as Dose Limiting Toxicities (DLT)
Description: Occurrence of any of the following toxicities, attributable to ENTO, during Cycle 1 was considered DLT:
  * Grade 4 non-hematologic toxicity except alopecia, nausea, and vomiting controllable with anti-emetic therapy, line associated venous thrombosis, infection-related toxicities such as fever/sepsis, and fatigue.
  * In participants without bone marrow evidence of hematologic malignancy, hematologic toxicity defined as failure to recover absolute neutrophil count (ANC > 500/μL) or platelet count (>25000/μL) within 28 days
  * Grade 4, clinically significant, electrolyte abnormalities that were not correctable within 24 hours
  * Liver function test abnormalities that did not resolve to Grade 2 within 10 days
  * Infection that resulted from unexpectedly complicated prolonged myelosuppression
  * Toxicities that required temporary interruption of treatment and did not resolve to Grade 2 within 10 days or ENTO was suspended or dose reduced for a period of more than 10 days.
Time Frame: Cycle 1 (28-day cycle)
Population: The DLT Analysis Set included all participants in the Full Analysis Set (all participants who received at least 1 dose of study drug [ENTO]) who received at least 21 days of ENTO or experienced a DLT during DLT assessment window.
Measure: Number; unit: percentage of participants
Arm/Group | ENTO 400 mg
Number analyzed (Participants) | 6
percentage of participants | 0.0

2. Secondary Outcome: Percentage of Participants With AEs and Laboratory Abnormalities Not Defined as DLT
Time Frame: Day 1 Up to 30 days after permanent discontinuation of study treatment (maximum approximately 80 weeks)
Population: Full Analysis Set included all participants who received at least 1 dose of study drug (ENTO).
Measure: Number; unit: percentage of participants
Arm/Group | ENTO 400 mg
Number analyzed (Participants) | 9
percentage of participants | 100.0

3. Secondary Outcome: Plasma Concentration of ENTO
Description: Plasma concentration of drug (ENTO) over different time points is reported.
Time Frame: Cycle 1 (28-days cycle) Day 8 at 0 (predose), 1, 2, 3, 4, 6, 8, and 12 hours postdose
Population: Pharmacokinetic (PK) Analysis Set included all participants in the Full Analysis Set who had necessary baseline and at least 1 non-missing post-treatment assessments. Participants with available data were analyzed. PK parameters were not derived from the collected data due to the early study termination.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ENTO 400 mg
Number analyzed (Participants) | 7
ng/mL
  Cycle 1 Day 8, predose | 921.9 (610.47)
  Cycle 1 Day 8, 1 hour postdose | 1395.7 (1081.40)
  Cycle 1 Day 8, 2 hours postdose | 1892.7 (1285.08)
  Cycle 1 Day 8, 3 hours postdose | 1529.1 (994.69)
  Cycle 1 Day 8, 4 hours postdose | 1350.0 (862.21)
  Cycle 1 Day 8, 6 hours postdose | 1139.3 (709.22)
  Cycle 1 Day 8, 8 hours postdose | 1075.9 (659.08)
  Cycle 1 Day 8, 12 hours postdose | 855.1 (568.18)

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days after permanent discontinuation of study treatment (maximum approximately 80 weeks)
Description: Full Analysis Set included all participants who received at least 1 dose of study drug (ENTO).
Arm/Group | ENTO 400 mg
All-Cause Mortality (participants affected / at risk) | 6/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ENTO 400 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1
Cataract (Eye disorders) | 1
Choroidal haemorrhage (Eye disorders) | 1
Pyrexia (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Hyphaema (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ENTO 400 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to sponsor's decision based on the results from the Phase 1b/2 Study GS-US-339-1559 (NCT02343939) in participants with Acute Myeloid Leukemia and reorganization of the drug development portfolio.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT03135028/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03135028/SAP_001.pdf